CLINICAL TRIAL: NCT03931252
Title: Thermic Effect of Feeding in Cystic Fibrosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HM20015037
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fat (Experimental): Boost VHC (Very High Calorie), Nestle, 8 ounce can
  Interventions: Dietary Supplement: Boost VHC
- High protein (Experimental): Ensure High Protein 8 ounce can
  Interventions: Dietary Supplement: Ensure High Protein

INTERVENTIONS:
Dietary Supplement: Boost VHC — 8 ounce can liquid meal, calories 530kcal, Carbohydrate 46g, Protein 22g, Fat 30g
  Arms: High fat
Dietary Supplement: Ensure High Protein — 8 ounce can liquid meal, calories 160kcal, Carbohydrate 13g, Protein 16g, Fat 2g
  Arms: High protein

SUMMARY:
The investigators propose to assess the contributions of the thermic effect of food intake (TEF), which is the amount of energy expended to digest food, to overall energy expenditure in Cystic Fibrosis (CF).

DETAILED DESCRIPTION:
Total energy expenditure (TEE) is comprised of the following components: resting energy expenditure (REE), thermic effect of food intake (TEF), adaptive thermogenesis (AT). The thermic effect of food is the amount of energy expended to digest food, and can be affected by factors such as protein / fat / carbohydrate contents of meals or the amount of time over which a meal is consumed. The investigators propose to assess the contributions of the thermic effect of food intake (TEF), which is the amount of energy expended to digest food, to overall energy expenditure in CF. Participants will be assigned to either a high fat liquid meal or a high protein liquid meal and assessed for components of energy expenditure in the whole room indirect calorimeter (metabolic chamber); participants will then be crossed over to the alternate liquid meal type, and differences in resting and total energy expenditure and the thermic effect of food will be assessed between the two types of meals.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of cystic fibrosis by Cystic Fibrosis Foundation-established criteria
* being followed at the VCU (Virginia Commonwealth University) Adult Cystic Fibrosis Center
* pulmonary and overall health status at baseline as assessed by pulmonary function testing and screening labs (complete blood count, liver enzymes, cholesterol, HgA1c). Criteria for baseline status are established for each individual patient as part of routine CF pulmonary care.
* ability to understand the study procedures and to comply with them for the entire length of the study

Exclusion Criteria:

* experiencing any signs or symptoms consistent with a pulmonary exacerbation (a decline in pulmonary function testing from baseline, recorded as part of routine CF care)
* undergoing treatment for a pulmonary exacerbation with a change in antibiotics or steroids from their baseline medications
* tobacco users
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Energy Expenditure | 16 hours after entry into metabolic chamber
  The changes in energy expenditure measured in kcal (resting energy expenditure prior to feeding, and thermic effect of food after meal administration) will be recorded in the metabolic chamber.

SECONDARY OUTCOMES:
glucose | 16 hours after entry into metabolic chamber
  blood glucose (mg/dL) measured with continuous glucose sensor and fasting venous sample at end of study visit
insulin | 16 hours after entry into metabolic chamber
  fasting insulin level (mIU/mL) measured at end of overnight visit
Leptin | 16 hours after entry into metabolic chamber
  fasting leptin level (ng/mL) measured at end of overnight visit
Ghrelin | 16 hours after entry into metabolic chamber
  fasting grehlin levels (pg/mL) measured at end of overnight visit

CONTACTS AND LOCATIONS:
Overall Officials: Trang Le, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No